CLINICAL TRIAL: NCT02617862
Title: The Use of the PCI Wide Field Imaging System for Pediatric Ophthalmic Photography of the Posterior and Peripheral Retina
Brief Title: PCI Imaging System in Pediatric Ophthalmology
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Proposed comparison (RetCam vs. COSMOS) was unfeasible. Device is now licensed in Canada.
Sponsor: Brenda Gallie (Other)
Collaborators: Phoenix Clinical Inc. (Industry)
Responsible Party: Sponsor-Investigator, Brenda Gallie, Ophthalmologist, The Hospital for Sick Children
Organization: The Hospital for Sick Children (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Sickkids
Record Dates: First submitted 2015-11-05; First posted 2015-12-01 (Estimated); Last update posted 2018-02-12 (Actual); Status verified 2018-02

CONDITIONS: Retinoblastoma
Keywords: Diagnostic imaging; Retina; Pediatrics
MeSH Terms: conditions — Retinoblastoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PCI imaging system (Experimental)
  Interventions: Procedure: Examination under anaesthetic (EUA); Device: RetCam; Device: COSMOS

INTERVENTIONS:
Procedure: Examination under anaesthetic (EUA) — The EUA is scheduled as part of the routine clinical management of children with various ophthalmic conditions.
Device: RetCam — The RetCam is a pediatric wide-field retinal camera that has been the mainstay for pediatric ophthalmic imaging since 1997. Imaging using the RetCam (during the EUA) is conducted as part of routine clinical magagement.
Device: COSMOS — The COSMOS images will be captured (during the EUA) after the RetCam images. The COSMOS is designed to be used in the same way as the RetCam, but to produce higher quality images.

SUMMARY:
The purpose of this study is to compare the RetCam (Clarity Medical Systems, Pleasanton, CA) to a new prototype pediatric imaging system, COSMOS, produced by Phoenix Clinical Incorporated (PCI) (Pleasanton, CA).

ELIGIBILITY:
* Exclusion Criteria:

  * Any patient who has a cloudy cornea.
  * Any patient whose RetCam imaging exam easily produces blanching of the optic nerve in the normal course of imaging.
  * Any patient who has consented to the procedure, but whose course of examination has filled the time allotted, leaving no time to evaluate the COSMOS.
* Inclusion Criteria:

  * Current patients undergoing clinically indicated EUA and RetCam imaging for surveillance and treatment of ophthalmic conditions at The Hospital for Sick Children.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2015-10; Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Comparison of the field of view in RetCam and COSMOS images | 1 day
  Masked investigators will review images from the RetCam and the COSMOS. Field of view will be graded on a scale from 1-5, with 1 being the worst and 5 being the best. We will test for significant difference, at alpha level 0.05, between scores of the images taken by the RetCam and the COSMOS.
Comparison of the color in RetCam and COSMOS images | 1 day
  Masked investigators will review images from the RetCam and the COSMOS. Color will be graded on a scale from 1-5, with 1 being the worst and 5 being the best. We will test for significant difference, at alpha level 0.05, between scores of the images taken by the RetCam and the COSMOS.
Comparison of the dynamic range in RetCam and COSMOS images | 1 day
  Masked investigators will review images from the RetCam and the COSMOS. Dynamic range will be graded on a scale from 1-5, with 1 being the worst and 5 being the best. We will test for significant difference, at alpha level 0.05, between scores of the images taken by the RetCam and the COSMOS.
Comparison of the sharpness in RetCam and COSMOS images | 1 day
  Masked investigators will compare images from the RetCam and the COSMOS and grade sharpness on a scale from 1-5, with 1 being the worst and 5 being the best. We will test for significant difference, at alpha level 0.05, between scores of the images taken by the RetCam and the COSMOS.
Comparison of the detail in RetCam and COSMOS images | 1 day
  Masked investigators will review images from the RetCam and the COSMOS. Detail will be graded on a scale from 1-5, with 1 being the worst and 5 being the best. We will test for significant difference, at alpha level 0.05, between scores of the images taken by the RetCam and the COSMOS.
Comparison of the resolution in RetCam and COSMOS images | 1 day
  Masked investigators will review images from the RetCam and the COSMOS. Resolution will be graded on a scale from 1-5, with 1 being the worst and 5 being the best. We will test for significant difference, at alpha level 0.05, between scores of the images taken by the RetCam and the COSMOS.
Comparison of the evenness of illumination in RetCam and COSMOS images | 1 day
  Masked investigators will review images from the RetCam and the COSMOS. Evenness of illumination will be graded on a scale from 1-5, with 1 being the worst and 5 being the best. We will test for significant difference, at alpha level 0.05, between scores of the images taken by the RetCam and the COSMOS.

CONTACTS AND LOCATIONS:
Overall Officials: Brenda L Gallie, MD, FRCSC, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada